CLINICAL TRIAL: NCT05060809
Title: Vitamin k Status and Its Relation to Vascular Calcification in Hemodialysis Patients in Assiut University Hospital
Brief Title: Vitamin k1 and Its Relation to Vascular Calcification in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshaimaa Sayed Hassan Mubarak, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: vit k in hemodialysis patient
Record Dates: First submitted 2021-09-19; First posted 2021-09-29 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Vascular Calcification
Keywords: hemodialysis; Vitamin k1
MeSH Terms: conditions — Vascular Calcification | interventions — Vitamin K 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodialysis patient with high level of dp uc-MGP (Experimental): one hundred and twenty hemodialysis patients with high level of dephosphorylated uc-MGP received 5 mg of oral vitamin K1 (phylloquinone) three times /week for 6 months at the end of HD session. We measured the serum dephosphorylated- uncarboxylated matrix Gla protein (dp-ucMGP) 6 months after vitamin K1 supplementation. In addition, plain lateral abdominal x-ray was conducted prior to and after 6 months of vitamin K supplementation to assess lumbar aorta calcification. The extent of aortic calcification score (AAC) was assessed by Kauppila score.In addition, study patients were subjected to an echocardiography at baseline as well as 6 months post vitamin K1 supplementation. Echocardiography was performed by the same operator.
  Interventions: Drug: oral vitamin k1 (phylloquinone)

INTERVENTIONS:
Drug: oral vitamin k1 (phylloquinone) — The enrolled patients received 5 mg of oral vitamin K1 (phylloquinone) three times /week for 6 months at the end of HD session to ensure compliance. We measured the serum dephosphorylated- uncarboxylated matrix Gla protein (dp-ucMGP) before and 6 months after vitamin K1 supplementation. In addition, plain lateral abdominal x-ray was conducted prior to and after 6 months of vitamin K supplementation to assess lumbar aorta calcification. The extent of aortic calcification score (AAC) was assessed by a semi-quantitative grading system developed by Kauppila.

SUMMARY:
Vascular calcification (VC) represents one of the major complications associated with progressive renal impairment. Matrix Gla-protein (MGP) is a vitamin K-dependent protein that acts as a powerful inhibitor of vascular calcification. Despite this fact, it remains unknown whether supplementation with vitamin K can lead to reduction or reversal of vascular and heart valve calcification. Our study aims primarily to investigate the effect of intravenous vitamin K1 three times weekly for a total duration of 6 months on the serum levels of dephosphorylated-uncarboxylated MGP (dp-ucMGP) as well as aortic calcification score and severity of aortic and mitral valve lesions.

DETAILED DESCRIPTION:
Vascular calcification (VC) represents one of the major complications associated with progressive renal impairment. In addition, VC has been regarded as one of the major predictors of cardiovascular risk, the most common cause of mortality in chronic kidney disease patients (CKD).

65% of end-stage kidney disease (ESKD) patients on regular peritoneal dialysis (PD) and 80-85% of ESKD patients on regular hemodialysis (HD) showed coronary or aortic calcification. These calcifications were associated with the total time on dialysis, with a yearly-increase of vascular calcification by 15% . Traditional risk factors for vascular calcification include age, male gender, smoking, diabetes, hypertension, and dyslipidemia.

VC, the pathological deposition of mineral in the vascular system, can manifest as intimal, medial, or heart valve calcification. Whereas intimal calcification, taking place within atherosclerotic plaque in aorta and coronary arteries, indicates advanced atherosclerosis, media calcification, which is often found in patients with diabetes and/or CKD, is characterized by diffuse mineral deposition along elastic fibers in both low resistance elastic-type as well as high resistance muscle-type arteries. Calciphylaxis, or calcific uremic arteriolopathy, represents a special form of ectopic, extraosseous calcification, that is characteristically observed in CKD patients, particularly those with ESKD with additional secondary hyperparathyroidism or those receiving warfarin. A study on hemodialysis patients showed more than two-fold higher odds of aortic and iliac calcifications in patients receiving warfarin than those who do not . VC results from an imbalance of promoters and inhibitors. Matrix Gla-protein (MGP) is a vitamin K-dependent protein and has been found to be expressed by medial vascular smooth muscles of arteries, endothelial cells, chondroblasts, and fibroblasts. Moreover, it is also expressed in the heart, kidneys, and lungs . MGP acts as a powerful inhibitor of vascular calcification. Loss-of-function mutations of MGP was associated with vascular calcification in animal models. In the setting of progressive vascular calcification, MGP transcription increases, giving rise to dephosphorylated-uncarboxylated MGP (dp-ucMGP). This molecule represents the inactive form of MGP, which later undergoes a γ- glutamate carboxylation and serine phosphorylation to produce the active form, phosphorylated carboxylated MGP (p- cMGP). Vitamin K acts as a cofactor for the enzyme γ-glutamylcarboxylase that is responsible for activating dp-ucGMP into dp-cMGP. Despite its key role in activation of dp-ucMGP, it remains unknown whether supplementation with vitamin K can lead to reduction or reversal of vascular and heart valve calcification in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥18 years of age,
* Not less than 6 months on HD,
* High level of serum dephosphorylated uc-MGP
* Signed informed consent,

Exclusion Criteria:

* Patients with normal level of dp-ucMGP
* History of thrombosis,
* Intake of vitamin K antagonists (warfarin) at baseline or in the 3 months prior to baseline,
* Inflammatory bowel disease,
* Liver dysfunction,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Effect of vitamin k1 supplementation on vascular calcification | 6 months
  Our study aims primarily to investigate the effect of oral vitamin K1 three times weekly for a total duration of 6 months on the serum levels of dephosphorylated-uncarboxylated MGP (dp-ucMGP) as well as aortic calcification score and severity of aortic and mitral valve lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Aoun M, Makki M, Azar H, Matta H, Chelala DN. High Dephosphorylated-Uncarboxylated MGP in Hemodialysis patients: risk factors and response to vitamin K2, A pre-post intervention clinical trial. BMC Nephrol. 2017 Jun 7;18(1):191. doi: 10.1186/s12882-017-0609-3. PMID 28592319
- [Background] Krueger T, Schlieper G, Schurgers L, Cornelis T, Cozzolino M, Jacobi J, Jadoul M, Ketteler M, Rump LC, Stenvinkel P, Westenfeld R, Wiecek A, Reinartz S, Hilgers RD, Floege J. Vitamin K1 to slow vascular calcification in haemodialysis patients (VitaVasK trial): a rationale and study protocol. Nephrol Dial Transplant. 2014 Sep;29(9):1633-8. doi: 10.1093/ndt/gft459. Epub 2013 Nov 26. PMID 24285427